CLINICAL TRIAL: NCT04595006
Title: Brown Fat Activation and Browning Efficiency Augmented by Chronic Cold and Nutraceuticals for Brown Adipose Tissue-mediated Effect Against Metabolic Syndrome (BEACON BEAMS Study)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Collaborators: Duke-NUS Graduate Medical School (Other); Canadian Imaging Research Centre (CIRC) (Other); National University of Singapore (Other); Singapore Institute of Food and Biotechnology Innovation (SIFBI) (Unknown); Singapore Bioimaging Consortium (SBIC) (Industry)
Responsible Party: Principal Investigator, Melvin Leow, Principal Investigator, Institute for Human Development and Potential (IHDP), Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018/00823
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Energy Expenditure; Obesity; Brown Adipose Tissue
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cold Stimulation (CS) (Experimental): Subjects will undergo a mild cold stimulation of about 14 degrees Celsius by wearing a cooling vest for approximately an hour daily for the next 12 weeks or 3 months.
  Interventions: Other: Cold Stimulation (CS)
- Browning Nutraceutical (BN) (Experimental): Subjects will consume 2000mg of curcumin daily for the next 12 weeks or 3 months.
  Interventions: Other: Browning Nutraceutical (BN)
- Cold Stimulation and Browning Nutraceutical (CSBN) (Experimental): Subjects will undergo a mild cold stimulation of about 14 degrees Celsius by wearing a cooling vest for approximately an hour and consume 2000mg of curcumin daily for the next 12 weeks or 3 months.
  Interventions: Other: Cold Stimulation and Browning Nutraceutical (CSBN)

INTERVENTIONS:
Other: Cold Stimulation (CS) — Subject wear cooling vest to stay cool
  Arms: Cold Stimulation (CS)
Other: Browning Nutraceutical (BN) — Subject will consume 2000mg of curcumin a naturally-occurring polyphenol antioxidant that is found in turmeric ginger rhizome root
  Arms: Browning Nutraceutical (BN)
Other: Cold Stimulation and Browning Nutraceutical (CSBN) — Subject wear a cooling vest and consume 2000mg of curcumin
  Arms: Cold Stimulation and Browning Nutraceutical (CSBN)

SUMMARY:
Our body fat (adipose tissue) is largely made up of white adipose tissue (WAT) that stores surplus energy as white fat depots. In addition, adult humans have another type of fat similar to the brown fat in babies that burns up fat to generate heat for maintenance of body temperature during cold exposure. Adults have much lesser amounts of such brown adipose tissue (BAT), most of which are located within the sides of the neck and under the skin above the collar bones as well as along the sides of the spine. BAT consists of both classical brown fat identical to that found in babies as well as beige fat (composed of brown-in-white or 'brite' fat cells) found mainly in adults. Both types of BAT burn fat upon activation by various stimuli such as cold or by substances like curcumin found in turmeric ginger rhizome root.

This study is carried out to find out the effects of cold stimulation and/or a known BAT-activating nutraceutical among those overweight/obese people suffering from metabolic syndrome.

DETAILED DESCRIPTION:
This study will recruit 60 participants that are overweight/obese people suffering from metabolic syndrome. The participants will be asked to come to the Clinical Nutrition Research Centre (CNRC) for a screening session (1st visit) and given plenty of time to read this information sheet and the opportunity to ask questions. Once the participants are fully informed regarding the study and all their questions have been satisfactorily answered, the participants will be given a consent form to complete and sign in the presence of the researcher. Following this, in order to gauge their suitability for taking part in the study, an assessment will be carried out. This assessment needs to be carried out in a fasted state and participants would therefore have to come one morning following an overnight fast. The screening will include anthropometric measurements, blood pressure measurement and blood sampling. Anthropometric measurements taken will be height, weight, waist circumference and hip circumference. Body composition will be measured using an electrical impedance analyser (BIA). Blood pressure will be measured using an automatic blood pressure monitor. The participants will also undergo a blood sampling from their vein (6 mL or approximately 1.5 teaspoons) to be tested for thyroid function, glucose and lipid profile. Pre-menopausal females will also undergo a urine pregnancy test to exclude pregnancy prior to participation at study entry. The participants who have been accepted into the study will be randomly assigned to one of the 3 parallel intervention groups below (20 subjects per group) via an online randomizer (www.randomizer.org). Randomization means assigning them to one of the three groups by chance, like tossing a coin or rolling a dice. The 3 parallel intervention groups (Week 0 to 12) are Group 1 (CS): Cold stimulation using cooling vest x 60 min once daily over 3 months, Group 2 (BN): Browning nutraceutical (2000mg curcumin) to be taken once daily over 3 months, Group 3 (CSBN): Cold stimulation using cooling vest x 60 min once daily and Browning nutraceutical (2000mg curcumin) to be taken once daily over 3 months. The participants will then be expected to come to the centre for a total of six separate test sessions, over a span of 6 months (2 test sessions each at week 0, 12 and 24 approximately +/-2 weeks). For each of the six test sessions,the participants will be required to fast overnight and avoid caffeine and alcohol for 8-10 hours, only plain water can be consumed during the fast before reporting at the CNRC in the morning between 8 to 9 am. The participants are to avoid any physical activity/exercise and alcohol on the day prior to the visit. The test sessions will be as follows: On the 2nd visit (first test session) at week 0, the participants will need come to CNRC in the morning and a fasting blood sample (40 mL or approximately 8 teaspoons) and urine sample will be collected before they undergo metabolic rate measurement with IRT focusing on their neck and area above the collar bone in a whole body room calorimeter for the next 45 minutes. The participants will then undergo a mild cold stimulation of about 14 degree Celsius by wearing a cooling vest for the next 45 minutes, in which metabolic rate measurement and IRT in the whole body calorimeter will be performed during this period. Please note that wearing the cooling vest may lead to some shivering, but it is generally considered safe. Upon exiting the whole body calorimeter, the participants will remove the cooling vest and then proceed to Clinical Imaging Research Centre (CIRC) located at the basement level of the same building, where an intravenous indwelling cannula will be inserted into an arm vein and 20 mL (approximately 4 teaspoons) of blood and another urine sample will be collected again. The participants will then wear the cooling vest again for approximately another 60 min and in between they will receive an intravenous injection of a radioactive labeled glucose called 18-FDG through the intravenous cannula. The cooling vest will be removed just prior to the start of the PET (Positron Emission Tomography) and MRI/MRS (Magnetic Resonance Imaging/Magnetic Resonance Spectroscopy) that will take place over the next 1 hour to quantify BAT (Brown Adipose Tissue) and abdominal white fat including liver and muscle fat. The participants will also need to undergo a body composition evaluation using dual energy X-ray absorptiometry (DXA) (approximately 20 mins duration) which allows quantification of fat, lean and bone mass. However, the participants will be given the option to do the DXA scan on their next/3rd visit according to their preference. After which, the participants will be free to leave. On the 3rd visit (second test session) at week 0, the participants will need come to CNRC in the morning for an Oral Glucose Tolerance Test (OGTT). Anthropometric measurements taken will be height, weight, waist circumference and hip circumference. Body composition will be measured using an electrical impedance analyser (BIA). Blood pressure will be measured using an automatic blood pressure monitor. A fasting blood sample (4 mL or less than 1 teaspoon) will be collected and participants will then be required to consume a glucose drink (75g of glucose) within 5 minutes. Subsequently after 120 min, another blood sample (4 mL or less than 1 teaspoon) will be collected. During the entire test session, the participants will have to stay rested and in the laboratory. Television and a workspace will be provided for the participants use if required. At the end of 2 hours of testing, for participants who have not undergone for the DXA scan on the 2nd visit, they will then proceed to complete the DXA scan (approximately 20 mins duration). After which, participants will be free to leave.The above 2 test sessions may be scheduled in any order,but to be completed no more than 2 weeks apart. The participants will now start the study intervention procedures as per the intervention group randomly assigned to them for the next 12 weeks or 3 months. Participants who are assigned to group 1 / cold stimulation (CS), will be expected to undergo a mild cold stimulation of about 14 degree Celsius by wearing a cooling vest for approximately an hour daily for the next 12 weeks or 3 months. Participants who are assigned to group 2 / browning nutraceutical (BN), will be expected to consume 2000mg of curcumin (in forms of capsules) daily for the next 12 weeks or 3 months. Curcumin is a naturally-occurring polyphenol antioxidant that is found in turmeric ginger rhizome root and has been widely known in Asia to have health benefits. Since both substances are commonly consumed among Asians, it is relevant to study their combined chronic clinical effects on BAT. Use of curcumin to stimulate BAT is essentially safe as both are naturally occurring plant derived substances from Curcuma longa rhizome. It is generally recognised as safe for human consumption. The US FDA has approved curcumin as 'Generally Recognised as Safe' (GRAS) status and allows these to be taken as foods ingredients. Participants who are assigned to group 3 / cold stimulation and browning nutraceutical (CSBN), will be expected to undergo a mild cold stimulation of about 14 degree Celsius by wearing a cooling vest for approximately an hour and, consume 2000mg of curcumin (in forms of capsules) daily for the next 12 weeks or 3 months. The participants will then be required to come for the 4th visit (third test session) and 5th visit (fourth test session) at week 12 (after completing the 3 months of intervention), as per follows:

On the 4th visit (third test session) at week 12, participants will repeat the same procedures as per that of the 2nd visit (first test session). For the 5th visit (fourth test session) at week 12, participants will need to come to CNRC in the morning in a fasted state and proceed first to CIRC for a 30 min MRI/ MRS only scan of BAT/WAT to study the fat composition. Subsequent procedures will be same as that of the 3rd visit (second test session). After which, there will be no more intervention and participants will continue with their usual lifestyle and diet for the next 3 months (week 12 to 24).The participants will lastly be required to come for the 6th visit (fifth test session) and 7th visit (sixth test session) at week 24 (6 months from start of study), and repeat the same procedures as per that of the 2nd visit (first test session) and the 3rd visit (second test session) respectively. Notes: *The 2 test sessions each at week 0, 12 and 24 may be scheduled within 4 weeks from each time point. *The following test sessions will be scheduled no more than 4 weeks apart: o First and second test sessions for Week 0 (in any order) o Third and fourth test sessions for Week 12 (in any order) o Fifth and sixth test sessions for Week 24 (in any order)

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Chinese, Malay or Indian ethnicity
* Age between 21 to 50 years
* Able to give informed consent
* Body mass index (BMI) between 23 to 32 kg/m2
* Thyroid function test must be within the normal ranges
* Willing to avail yourself for the whole study and follow study procedures
* EITHER deemed to have pre-metabolic syndrome when waist circumference is > 90 cm in men or > 80 cm in women, with none or up to one of the following condition:

  * Triglyceride level ≥ 1.7 mmol/L
  * HDL cholesterol ≤ 1.0 mmol/L in men, and ≤ 1.3 mmol/L in women
  * Blood pressure ≥ 130/85 mmHg
  * Fasting blood glucose of ≥ 6.1 mmol/L
* OR deemed to have metabolic syndrome when three or more of the following conditions are present:

  * Waist circumference > 90 cm in men and > 80 cm in women
  * Triglyceride level ≥ 1.7 mmol/L
  * HDL cholesterol ≤ 1.0 mmol/L in men, and ≤ 1.3 mmol/L in women
  * Blood pressure ≥ 130/85 mmHg
  * Fasting blood glucose of ≥ 6.1 mmol/L

Exclusion Criteria:

* Are pregnant or contemplating pregnancy (for female subjects)
* Partake in sports at the competitive and/or endurance levels
* Have known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Have major chronic disease such as heart disease or cancer
* Take insulin or drugs known to affect glucose metabolism
* Intentionally restrict food intake
* Have major medical or surgical event requiring hospitalization within the preceding 3 months
* Have taken antibiotics for 3 months before the study period
* Are a smoker
* Are an overnight shift worker
* Have any known food allergy (eg. anaphylaxis to peanuts)
* Having active Tuberculosis (TB) or currently receiving treatment for TB
* Have any known Chronic Infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Are a member of the research team or their immediate family members. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Enrolled in a concurrent research study judged not to be scientifically or medically compatible with the study of the CNRC
* Have poor veins impeding venous access
* Have any history of severe vasovagal syncope (blackouts or near faints) following blood draws
* History of surgery with metallic clips, staples or stents
* Presence of cardiac pacemaker or other foreign body in any part of the body
* History of claustrophobia particularly in a MRI scanner

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2028-08-16 (Estimated)

PRIMARY OUTCOMES:
Change in Brown adipose tissue activation detection by Imaging using 18-FDG-PET/ MRI. | Week 0, 12 and 24 of cold stimulus
Change in Brown adipose tissue activation detection by Imaging using Infrared | Week 0, 12 and 24 of cold stimulus
Change in Energy Expenditure using Whole Body Calorimeter. | Week 0, 12 and 24 of cold stimulus
Change in Brown adipose tissue activation detection by Imaging using 18-FDG-PET/ MRI. | Week 0, 12 and 24 of consumption of Curcumin
Change in Brown adipose tissue activation detection by Imaging using Infrared | Week 0, 12 and 24 of consumption of Curcumin
Change in Energy Expenditure using Whole Body Calorimeter. | Week 0, 12 and 24 of consumption of Curcumin
Change in Brown adipose tissue activation detection by Imaging using 18-FDG-PET/ MRI. | Week 0, 12 and 24 of cold stimulus and consumption of curcumin
Change in Brown adipose tissue activation detection by Imaging using Infrared | Week 0, 12 and 24 of cold stimulus and consumption of curcumin
Change in Energy Expenditure using Whole Body Calorimeter. | Week 0, 12 and 24 of cold stimulus and consumption of curcumin

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore Institute of Clinical Sciences, Singapore, Singapore